CLINICAL TRIAL: NCT06768333
Title: The Need for Speed: Comparing the Speed of Glucose Absorption During Repeated Sprint Cycling
Brief Title: Speed of Glucose Absorption During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster University (Other)
Responsible Party: Principal Investigator, Dr. Chris Gaffney, Principal Investigator, Lancaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LMS-24-Dean-2
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-01

CONDITIONS: Healthy Nutrition; Healthy

STUDY DESIGN:
Intervention Model Description: This will be a double-blind randomised crossover design. There will be 1 group of participants who will complete all three conditions at random:
  Condition 1 - consume Voom Pocket Rocket. Condition 2 - consume SIS Isotonic Energy Gel. Condition 3 - consume Maurten Gel 160.
  Participants will consume each product 35 minutes before starting exercise.
  All participants will undergo the same exercise - 5 repeated sprint cycling (cycling against 0.075 kg/ kg body mass) intervals of 15 seconds interspersed with 3 minutes of active recovery.
  All participants will have the same measures taken - blood sampling for blood glucose, blood lactate, and electrolytes at the end of each sprint and period of active recovery, and monitoring of gas exchange throughout the exercise.
Who Masked: Participant, Investigator
Masking Description: Both the participants and investigators will be blinded to what supplement they are consuming on each visit. Each supplement will taste the same, and be placed into identical packaging, and be randomly labelled (e.g., A, B, C). This will be done to avoid potential bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Voom Pocket Rocket Electro Energy Bar (Experimental): After at least 48 hours, every participant will undergo a different condition
  Interventions: Dietary Supplement: 45 grams Voom Pocket Rocket Electro Energy
- Maurten Gel 160 (Experimental): After at least 48 hours, every participant will undergo a different condition
  Interventions: Dietary Supplement: 45 grams Maurten Gel 160
- SIS Go Isotonic Energy Gel (Experimental): After at least 48 hours, every participant will undergo a different condition
  Interventions: Dietary Supplement: 45 grams SIS Go Isotonic Energy Gel

INTERVENTIONS:
Dietary Supplement: 45 grams Voom Pocket Rocket Electro Energy — Participants will be required to consume 45 grams (in carbohydrates) of the Voom Pocket Rocket Electro Energy on one of the three experimental visits. Participants will have blood glucose, blood lactate, and electrolytes sampled throughout five 15-second repeated cycling intervals interspersed with 3 minutes active recovery. Gas exchange will also be monitored throughout the 1-hour study visit.
  Arms: Voom Pocket Rocket Electro Energy Bar
Dietary Supplement: 45 grams Maurten Gel 160 — Participants will be required to consume 45 grams (in carbohydrates) of the Maurten Gel 160 on one of the three experimental visits. Participants will have blood glucose, blood lactate, and electrolytes sampled throughout five 15-second repeated cycling intervals interspersed with 3 minutes active recovery. Gas exchange will also be monitored throughout the 1-hour study visit.
  Arms: Maurten Gel 160
Dietary Supplement: 45 grams SIS Go Isotonic Energy Gel — Participants will be required to consume 45 grams (in carbohydrates) of the SIS Go Isotonic Energy Gel on one of the three experimental visits. Participants will have blood glucose, blood lactate, and electrolytes sampled throughout five 15-second repeated cycling intervals interspersed with 3 minutes active recovery. Gas exchange will also be monitored throughout the 1-hour study visit.
  Arms: SIS Go Isotonic Energy Gel

SUMMARY:
The purpose of this study is to look at how fast commercially available supplements containing carbohydrates can get into the bloodstream during repeated sprint cycles. This will build from a pervious study where the investigators tested these supplements on healthy participants during a resting oral glucose tolerance trial. The investigators will be testing three supplements, namely Voom Pocket Rocket, SIS Go Isotonic Energy Gel, and Maurten Gel 160. Each participant will complete all three conditions, consuming one of each supplement at random per condition. The study requires participation from male and female runners, cyclists and triathletes who are aged between 18-40.

Each visit will take approximately 1 hour, and three experimental visits per participant. The study will involve frequent blood sampling and the continuous monitoring of gas exchange (oxygen/carbon dioxide). Blood sampling via cannulation will be used to analyse the lactate, glucose, and electrolyte content of the blood. Gas exchange will measure the oxygen breathed in and carbon dioxide breathed out throughout the exercise.

The investigators plan to carry out the study on 10 participants who will be a mix of male and female runners, cyclists and triathletes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-40 years
* Male or female
* Tier 2 athletes - local level representation, training ~ 3 times per week, training with a purpose to compete, identify with a specific sport, limited skill development (McKay et al., 2021)

Exclusion Criteria:

* Allergies to any listed ingredients on any supplements.
* Diabetes (type 1 or 2)
* Any medical conditions
* Smokers
* Any injury that would prevent them from exercising
* Anyone using drugs or medication (not including contraception)
* Anyone consuming alcohol within 24 hours of the study
* Exercise must be restricted within 24 hours of the study
* Caffeine must not be consumed within 24 hours of testing as it can significantly enhance carbohydrate oxidation rates (Yeo et al., 2005)
* Diets including high-carbohydrate-low-fat (HCLF), low-carbohydrate-high-fat (LCHF), ketogenic, and/or glycogen manipulation diets (Rauch et al., 2022)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males and Females
Enrollment: 10 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | Blood glucose measures will be taken 35 minutes after consuming the supplement(s) (baseline), after the 3 minute warmup, and then after every 15 second sprint and every 3 minute period of active recovery
  Frequent blood sampling for blood glucose (1ml after every stage of both sprint cycling and active recovery) followed by analysis in the Biosen Analyser
Blood Lactate | Blood lactate measures will be taken 35 minutes after consuming the supplement(s) (baseline), after the 3 minute warmup, and then after every 15 second sprint and every 3 minute period of active recovery
  Frequent blood sampling for blood lactate (1ml after every stage of both sprint cycling and active recovery) followed by analysis in the Biosen Analyser
Gas Exchange | Gas exchange will be measured continuously throughout the 20 minutes of exercise, starting at the warmup
  Gas exchange measured throughout each 20 minute exercise via a Cortex Metalyzer

SECONDARY OUTCOMES:
Blood electrolyte content | Blood electrolyte measures will be taken 35 minutes after consuming the supplement(s) (baseline), after the 3 minute warmup, and then after every 15 second sprint and every 3 minute period of active recovery
  Frequent blood sampling for electrolyte concentrations of the blood (sodium, potassium, chloride, calcium) (1ml after every stage of both sprint cycling and active recovery) followed by analysis in the Biosen Analyser
Rate of Percieved exertion (RPE) | RPE will be measured at the end of the warmup and the end of the final sprint stage
  Participants will report their RPE using the Borg Scale to report how hard they are finding the exercise. This will be done after the warm-up and after the final sprint.
Gastrointestinal (GI) Discomfort Questionnaire | GI Discomfort will be measured 5 minutes before and 5 minutes after exercise
  Participants will complete a GI discomfort questionnaire 5 minutes before starting exercise and at the end of exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Lancaster University, Lancaster, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rauch CE, McCubbin AJ, Gaskell SK, Costa RJS. Feeding Tolerance, Glucose Availability, and Whole-Body Total Carbohydrate and Fat Oxidation in Male Endurance and Ultra-Endurance Runners in Response to Prolonged Exercise, Consuming a Habitual Mixed Macronutrient Diet and Carbohydrate Feeding During Exercise. Front Physiol. 2022 Jan 4;12:773054. doi: 10.3389/fphys.2021.773054. eCollection 2021. PMID 35058795